CLINICAL TRIAL: NCT03862755
Title: Chemoprophylaxis Plus Early Ambulation Prevent Chinese Thoracic Surgery Patients From Pulmonary Embolism
Brief Title: Chemoprophylaxis Plus Early Ambulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shen Lei (Other)
Responsible Party: Sponsor-Investigator, Shen Lei, Clinical Associated Professor, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PE Prevention in SPH
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Embolism; Thoracic Surgery
Keywords: Pulmonary embolism; Thoracic surgery; Thromboprophylaxis
MeSH Terms: conditions — Pulmonary Embolism | interventions — Chemoprevention; Heparin, Low-Molecular-Weight; Early Ambulation

STUDY DESIGN:
Intervention Model Description: Early chemoprophylaxis means low-molecular weight heparin (LMWH) 3075 IU (WHO Units) injection subcutaneously one time a day no later than 24 hours after surgery. Early ambulation means activity out of bed no later than 24 hours after surgery. According to different risk level, patients received different thromboprophylaxis strategies. Early ambulation alone was for patients at low risk (Caprini 0-4), early chemoprophylaxis plus early ambulation was for patients at moderate (Caprini 5-8) or high risk (Caprini ≥9).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Thromboprophylaxis (Experimental): All surgical patients classified into low risk and moderate/high risk groups based on Caprini score and received different thromboprophylaxis strategies Briefly, early ambulation alone was used in patients at low risk, early ambulation plus chemoprophylaxis with Low Molecular Weight Heparin was used in patients at moderate/high risk.
  Interventions: Drug: Chemoprophylaxis with Low Molecular Weight Heparin (LMWH)

INTERVENTIONS:
Drug: Chemoprophylaxis with Low Molecular Weight Heparin (LMWH) — Early chemoprophylaxis means low-molecular weight heparin (LMWH) 3075 IU (WHO Units) injection subcutaneously one time a day no later than 24 hours after surgery. Early ambulation means activity out of bed no later than 24 hours after surgery. According to different risk level, patients received different thromboprophylaxis strategies. Early ambulation alone was for patients at low risk (Caprini 0-4), early chemoprophylaxis plus early ambulation was for patients at moderate (Caprini 5-8) or high risk (Caprini ≥9).
  Other Names: Early ambulation

SUMMARY:
Pulmonary embolism (PE) can be a devastating postoperative complication and the leading cause of mortality after thoracic surgery. PE together with deep venous thrombosis (DVT) is called venous thromboembolism (VTE), whereas PE caused much more serious situation than DVT. Huge amount of data have demonstrated that thromboprophylaxis after surgery is very important to prevent postoperative VTE, especially after orthopedic surgery and plaster surgery. Moreover, for thoracic surgery, American College of Chest Physicians (ACCP) has published prevention guidelines of VTE in non-orthopedic surgical patients and has been used widely, but unfortunately prophylaxis measures had often been underused in China. However, to be honest, there could be a big difference between Chinese and western populations, for example, what guidelines recommended thrombolysis therapy in diagnosed massive or sub-massive PE patients is tissue type plasminogen activator (t-PA) 100 mg, while in China 50 mg has the same effect. So investigators wanted to establish if the prophylaxis measures what they were using currently are suitable for Chinese thoracic surgical patients.

DETAILED DESCRIPTION:
Investigators enrolled 598 patients who were sent to thoracic postoperative intensive care unit (ICU) ward right after surgery from August 8 to September 12 of 2017 and those patients stayed in ICU for at least 24 hours. Excluded non-lung surgery there were 581 lung surgery cases. Investigators adopted the Caprini VTE risk assessment model from Boston Medical Center (BMC) in United States of America (USA). According to different risk level, participants received different thromboprophylaxis strategies. Early ambulation alone was for patients at low risk (Caprini 0-4), early chemoprophylaxis plus early ambulation was for patients at moderate (Caprini 5-8) or high risk (Caprini ≥9). Early chemoprophylaxis means low-molecular weight heparin (LMWH) 3075 IU (WHO Units) injection subcutaneously one time a day no later than 24 hours after surgery. Early ambulation means activity out of bed no later than 24 hours after surgery. Thromboprophylaxis contraindication included chest tube drainage more than 500 ml or major bleeding during operation or surgeons refusing to use thromboprophylaxis because they thought that patients would benefit more from not performing early ambulation or chemoprophylaxis. Some patients received chemoprophylaxis after they moved back to regular ward out of ICU which was called late chemoprophylaxis which means more than 24 hours after surgery. All chemoprophylaxis were used only during hospitalization. When participants were discharged, no extended treatment prescribed. However, they were followed up twice on 30 days and 60 days after surgery by phone call.

ELIGIBILITY:
Inclusion Criteria:

* Lung surgical patients who were sent to thoracic postoperative intensive care unit (ICU) ward right after surgery and stayed in ICU for at least 24 hours.

Exclusion Criteria:

* Cases received inferior vena filter and anti-coagulation treatment history.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gening Jiang, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Thromboprophylaxis: All surgical patients classified into low risk and moderate/high risk groups based on Caprini score and received different thromboprophylaxis strategies Briefly, early ambulation alone was used in patients at low risk, early ambulation plus chemoprophylaxis with Low Molecular Weight Heparin was used in patients at moderate/high risk.
  Chemoprophylaxis with Low Molecular Weight Heparin (LMWH): Early chemoprophylaxis means low-molecular weight heparin (LMWH) 3075 IU (WHO Units) injection subcutaneously QD no later than 24 hours after surgery. Early ambulation means activity out of bed no later than 24 hours after surgery. According to different risk level, patients received different thromboprophylaxis strategies. Early ambulation alone was for patients at low risk (Caprini 0-4), early chemoprophylaxis plus early ambulation was for patients at moderate (Caprini 5-8) or high risk (Caprini ≥9).
Period: Overall Study
Arm/Group | Thromboprophylaxis
Started | 581
Completed | 581
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 581
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 293
  Male | 288
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 581
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 23.3 (3.2)
Pathologic diagnosis [Number; unit: participants]
  Malignant | 433
  Benign | 148
Surgical procedure [Number; unit: participants]
  Sub-lobar resections | 188
  Lobectomy | 368
  Extended Lobectomy | 25
Length of ICU stay [Mean (Standard Deviation); unit: days] | 1.2 (0.6)
Length of Hospital Stay [Mean (Standard Deviation); unit: days] | 8.8 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Pulmonary Embolism (PE) in Surgical Thoracic Patients Under Currently Used PE Prevention Strategies.
Description: Real number of PE cases are recorded. PE cases are confirmed by computed tomographic pulmonary angiography (CTPA). During hospitalization, on postoperative 30 days and 60 days, PE incidence is recorded and compared with that of some retrospective patients group. Investigators will study if currently used prevention strategies are effective to prevent PE.
Time Frame: up to 8 weeks post operation
Measure: Count of Participants; unit: Participants
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 581
Participants | 3

2. Secondary Outcome: Provider Adherence in Implementation of PE Prevention Strategies.
Description: Since thromboprophylaxis is often underused in China, investigators want to investigate provider adherence in complying with thromboprophylaxis implementation. Some provider, mainly surgeon, don't comply with currently used prevention strategies. Based on real prevention methods that patients have received during postoperative period, provider adherence are shown as percentage. When analyzing data, investigators need to exclude those patients who didn't receive proper prevention according to our guidelines from whole patients group. By studying adherence outcome, investigators will know in what extent the surgeon's decision will influence the result.
Time Frame: Through study completion, an average of 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 581
Participants
  Compliance | 306
  Non-compliance | 275

ADVERSE EVENTS:
Time Frame: until 2 days from the last intake of LMWH, an average of 72 hours
Description: Major bleeding
Arm/Group | Thromboprophylaxis
All-Cause Mortality (participants affected / at risk) | 1/581
Serious Adverse Events (participants affected / at risk) | 0/581
Other Adverse Events (participants affected / at risk) | 0/581

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03862755/Prot_SAP_002.pdf